CLINICAL TRIAL: NCT02251158
Title: Relative Bioavailability of 500/200 mg of Tipranavir/Ritonavir Paediatric Solution Compared to 500/200 mg of Tipranavir/Ritonavir Capsules Following Oral Administration and Bioavailability of 500/200 mg Tipranavir/Ritonavir Paediatric Solution Under the Influence of Food in Healthy Female and Male Subjects. An Open-label, Randomised, Single-dose, Three-way Crossover Trial.
Brief Title: Bioavailability of Tipranavir/Ritonavir Paediatric Solution Compared to Tipranavir/Ritonavir Capsules in Healthy Female and Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1182.45
Record Dates: First submitted 2014-09-25; First posted 2014-09-29 (Estimated); Last update posted 2014-09-29 (Estimated); Status verified 2014-09

CONDITIONS: Healthy
MeSH Terms: interventions — tipranavir; Ritonavir

ARMS (3):
- TPV/r with food (Experimental): Tipranavir/Ritonavir paediatric/oral solution
  Interventions: Drug: Tipranavir oral solution; Drug: Ritonavir oral solution; Other: High fat breakfast
- TPV/r (Experimental): Tipranavir/Ritonavir paediatric/oral solution
  Interventions: Drug: Tipranavir oral solution; Drug: Ritonavir oral solution
- TPV/r capsules (Active Comparator)
  Interventions: Drug: Tipranavir capsules; Drug: Ritonavir soft gel capsules

INTERVENTIONS:
Drug: Tipranavir oral solution
  Arms: TPV/r; TPV/r with food
Drug: Tipranavir capsules
  Arms: TPV/r capsules
Drug: Ritonavir oral solution
  Arms: TPV/r; TPV/r with food
Drug: Ritonavir soft gel capsules
  Arms: TPV/r capsules
Other: High fat breakfast
  Arms: TPV/r with food

SUMMARY:
Study to determine the relative bioavailability of 500/200 mg of tipranavir/ritonavir (TPV/r) oral solution compared to 500/200 mg of TPV/r capsules following oral administration and to investigate the relative bioavailability of 500/200 mg of TPV/r oral solution with food versus without food.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and females according to the following criteria:

   Based upon a complete medical history, including the physical examination, vital signs (BP, HR), 12-lead ECG, clinical laboratory tests
   * No finding deviating from normal and of clinical relevance
   * No evidence of a clinically relevant concomitant disease
2. Age ≥ 18 and Age ≤ 55 years
3. BMI ≥ 18.5 and BMI ≤ 29.9 kg/m2 (Body Mass Index)
4. Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice and the local legislation

Exclusion Criteria:

1. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
2. Surgery of gastrointestinal tract (except appendectomy)
3. Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
4. History of relevant orthostatic hypotension, fainting spells or blackouts
5. Chronic or relevant acute infections
6. History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
7. Intake of drugs with a long half-life (>24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
8. Use of drugs which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial (e.g. drugs which contain polyethylene glycol or vitamin E)
9. Participation in another trial with an investigational drug within two months prior to administration or during the trial
10. Smoker (more than 10 cigarettes/day or 3 cigars/day or 3 pipes/day)
11. Inability to refrain from smoking on trial days
12. Alcohol abuse (more than 60 g/day)
13. Drug abuse
14. Veins unsuited for iv puncture on either arm (e.g. veins which are difficult to locate, access or puncture, veins with a tendency to rupture during or after puncture)
15. Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
16. History of any bleeding disorder or acute blood coagulation defect of vitamin K deficiency caused by anticoagulation therapy or malabsorption
17. Vitamin E supplement intake
18. Excessive physical activities (within one week prior to administration or during the trial)
19. Any laboratory value outside the reference range that is of clinical relevance
20. Inability to comply with dietary regimen of study centre

    For female subjects:
21. Pregnancy
22. Positive pregnancy test
23. No adequate contraception e.g. oral contraceptives, sterilization, intrauterine device
24. Inability to maintain this adequate contraception during the whole study period
25. Lactation period

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2003-10; Primary Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
AUC0-∞ (area under the concentration time curve of tipranavir in plasma over the time interval from 0 extrapolated to infinity) | up to 72 hours after drug administration
Cmax (maximum concentration of tipranavir in plasma) | up to 72 hours after drug administration

SECONDARY OUTCOMES:
AUC0-tz (area under the concentration-time curve of tipranavir in plasma over the time interval from 0 to the time of the last quantifiable data point) | up to 72 hours after drug administration
tmax (time from dosing to the maximum concentration of tipranavir in plasma) | up to 72 hours after drug administration
t1/2 (terminal half-life of tipranavir in plasma) | up to 72 hours after drug administration
MRTpo (mean residence time of the analyte in the body after oral administration) | up to 72 hours after drug administration
CLpo/F (apparent clearance of tipranavir in the plasma after extravascular administration) | up to 72 hours after drug administration
Vz/F (apparent volume of distribution during the terminal phase λz following an extravascular dose) | up to 72 hours after drug administration
Number of subjects with adverse events | up to day 18